CLINICAL TRIAL: NCT02380638
Title: Effects of Whole-body Vibration Training on Bone Mass and Bone Metabolism in Adolescents With Down Syndrome / Efectos Del Entrenamiento Vibratorio en la Masa ósea y el Metabolismo óseo de Adolescentes Con síndrome de Down
Brief Title: Effects of Whole-body Vibration Training on Body Composition in Adolescents With and Without Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, José A. Casajús, MD, PhD., Universidad de Zaragoza
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: DEP2009-09183
Record Dates: First submitted 2015-02-20; First posted 2015-03-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-02

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

ARMS (4):
- DS-WBV (Experimental): Exercise with Whole-body vibration (WBV) platform (Power Plate®). The participants will perform squat on a vibratory platform (3 times per week; 10 repetitions 30 to 60 seconds; Frequency: 25-30 Hz; Amplitude: 2 mm).
  Interventions: Device: Whole-body vibration training (Power Plate®) on bone mass and bone metabolism in adolescents with and without Down syndrome.
- DS-NONWBV (No Intervention): This group will continue with their day-to-day lifestyle during the course of the project.
- NONDS-WBV (Experimental): Exercise with Whole-body vibration (WBV) platform (Power Plate®). The participants will perform squat on a vibratory platform (3 times per week; 10 repetitions 30 to 60 seconds; Frequency: 25-30 Hz; Amplitude: 2 mm).
  Interventions: Device: Whole-body vibration training (Power Plate®) on bone mass and bone metabolism in adolescents with and without Down syndrome.
- NONDS-NONWBV (No Intervention): This group will continue with their day-to-day lifestyle during the course of the project.

INTERVENTIONS:
Device: Whole-body vibration training (Power Plate®) on bone mass and bone metabolism in adolescents with and without Down syndrome.
  Arms: DS-WBV; NONDS-WBV

SUMMARY:
The main aims of the present project include 1) to study the longitudinal effects of whole-body vibratory exercise on bone metabolism in adolescents with and without DS and 2) to evaluate whether a low frequency vibratory training program consisting of 3 sessions per week for 9 months (each vibratory session last approximately 10 minutes and includes 5-6 bouts of 1 min with 1 min rest between bouts) can improve bone development in these populations. Finally, and additional aim of the project is 3) to determine how long these effects may last after the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Both groups: Ages 10 - 19.
* Both groups: Parental/guardian permission (informed consent) and if appropriate, child verbal assent.
* Down syndrome group only: Diagnosis of Down syndrome.

Exclusion Criteria:

* Taking medication affecting bone.
* Non-caucasian.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2010-01; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in body composition assessed with dual energy X-ray at different time points, 6 months and 15 months. | Changes from baseline in body composition at 6 months and changes from baseline in body composition at 15 months

SECONDARY OUTCOMES:
Changes from baseline in bone structure evaluated with peripheral quantitative computed tomography at different time points, 6 months and 15 months. | Changes from baseline in bone structure at 6 months and changes from baseline in bone structure at 15 months

CONTACTS AND LOCATIONS:
Overall Officials: José A. Casajús, MD, PhD, Principal Investigator — GENUD Research Group
Locations (1):
- GENUD Research Group, Zaragoza, Zaragoza, Spain